CLINICAL TRIAL: NCT01409590
Title: Exercise and Diet Program for Schizophrenia Patients Who Are Taking Atypical Antipsychotic Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Revital Amiaz, MD, Sheba Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SHEBA-05-3627-RA-CTIL
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; weight gain; atypical neuroleptics
MeSH Terms: conditions — Schizophrenia; Weight Gain | interventions — Resistance Training; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise and Diet program (Other): All patients recruited in the study, participated in an homogeneous exercise program and diet.
  Interventions: Behavioral: Exercise program; Behavioral: Diet

INTERVENTIONS:
Behavioral: Exercise program — Homogenous exercise program in local fitness centers
Behavioral: Diet — Weigh loss diet program prescribed by a professional nutritionist

SUMMARY:
In this study the investigators will recruit patients with the diagnosis of schizophrenia that are taking atypical neuroleptics and that are willing to participate in an exercise and diet program. The investigators will measure weight and abdomen circumference.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia
* Atypical neuroleptics

Exclusion Criteria:

* Medical illness preventing exercise

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2005-05; Primary Completion 2006-09 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Weight loss | One year
  The weight of the participants of the trial was monitored during the trial, while they were following the exercise program and the diet, starting from the baseline until end of study/early withdrawal.

SECONDARY OUTCOMES:
Abdomen circumference | One year
  The circumference of the abdomen of the participants of the trial was monitored during the trial, while they were following the exercise program and the diet, starting from the baseline until end of study/early withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Revital Amiaz, MD, Principal Investigator — Sackler School of Medicine
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Ramat Gan, Israel